CLINICAL TRIAL: NCT00756262
Title: Probiotic Lactobacillus GG to Eliminate VRE Colonization
Acronym: VRE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment, no additional funding available
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6283; 5 R 21 AT-001892
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Vancomycin Resistant Enterococcal Colonization
Keywords: Vancomycin Resistant enterococcal colonization; Probiotics; LGG; Lactobacillus rhamnosus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lactobacillus rhamnosus LGG
  Interventions: Biological: Lactobacillus GG or Culturelle
- 2 (Placebo Comparator): Microcrystalline cellulose capsules
  Interventions: Biological: Lactobacillus GG or Culturelle

INTERVENTIONS:
Biological: Lactobacillus GG or Culturelle — Drug to be administered orally (capsule form). Dose=2 capsules/day for 14 days. Dosage strength= 1x10^10 bacteria
  Other Names: Lactobacillus GG (LGG); Placebo is microcrystalline cellulose

SUMMARY:
The use of LGG will be associated with elimination of VRE colonization.

The primary comparison will be VRE elimination rates among those patients that receive LGG compared to those that receive placebo. The primary endpoint will be the proportion of patients with VRE at one week after cessation of administration of study medication or placebo. The investigators assume that the placebo group will have very little spontaneous elimination of VRE and that the LGG group will be more likely to have eliminated VRE colonization at the end of one week.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Identified as having had a clinical isolate or stool or rectal swab culture positive for VRE
3. Able to give informed consent and report on side effects
4. Tolerating an oral/enteral diet
5. Stable comorbid conditions
6. Willing and able to come to Tufts for weekly visits
7. Outpatient

Exclusion Criteria:

1. Inpatients
2. Active infection with VRE being treated
3. Pregnancy
4. Known use of LGG or another probiotic (not including yogurt) within the previous 30 days
5. Presence of an active bowel leak, acute abdomen, active intestinal disease, or significant bowel dysfunction
6. Presence of an absolute neutrophil count less than 500 per cubic mm or anticipation post chemotherapy that the absolute neutrophil count will fall below 500 per cubic mm
7. History of adverse reaction to product containing lactobacillus
8. Active colitis (see definition below)
9. Treatment with an antibiotic with activity against VRE
10. Life expectancy less than one year or life-threatening condition
11. Known or suspected allergies to probiotics, lactobacillus, milk protein, and microcrystalline cellulose
12. Structural heart disease, history of endocarditis or valve replacement
13. Positive baseline stool culture for LGG
14. Recent or planned chemotherapy or radiation therapy
15. Solid organ transplant within the prior year
16. Stem cell transplant within the prior year
17. On active immunosuppressive medication [anti-rejection, injectable immunosuppressive drugs for autoimmune disease, or corticosteroids (greater than 1/2 mg per kg body weight of prednisone or its equivalent) not including inhaled or topical steroids]
18. Allergy or intolerance to or contraindication to two or more of the rescue antibiotic regimens (ampicillin, clindamycin, moxifloxacin)

Colitis will be defined as a history of Crohn's disease or ulcerative colitis with active diarrhea, active diarrhea due to Clostridium difficile infection, active diarrhea due to known or unknown cause with a stool specimen showing fecal leukocytes (if none has been done in such a patient this will be requested prior to enrollment). Diarrhea will be defined as more than three unformed bowel movements per day. The subject's primary physician will be asked to assess the subject's life expectancy, and subjects with an estimated life expectancy of less than one year as judged by the physician who knows him or her best will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the proportion of patients with VRE at one week after cessation of administration of study medication or placebo. | Day 21post enrollment

SECONDARY OUTCOMES:
The rate of VRE colonization in LGG recipients versus controls at 2 weeks and 6 weeks post discontinuation of administration of LGG or placebo. | 2 weeks, and 6 weeks
The rate of LGG colonization in study population receiving LGG compared to placebo. | days 21, 28, 56
That LGG can be used safely and without significant side effects in both hospitalized and ambulatory patients. | day 0-56 and 6 mnths
That among those treated with LGG, the colony counts of VRE will be lower when compared to controls even among those in whom colonization is not eliminated. | day 0,7,14,21,28,56

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center-Division of Geographic Medicine and Infectious Diseases, Boston, Massachusetts, United States

REFERENCES:
- [Result] Doron S, Hibberd PL, Goldin B, Thorpe C, McDermott L, Snydman DR. Effect of Lactobacillus rhamnosus GG Administration on Vancomycin-Resistant Enterococcus Colonization in Adults with Comorbidities. Antimicrob Agents Chemother. 2015 Aug;59(8):4593-9. doi: 10.1128/AAC.00300-15. Epub 2015 May 26. PMID 26014940